CLINICAL TRIAL: NCT00003105
Title: Phase I/II Trial of Sequential Doxorubicin/Gemcitabine (AG) and Ifosfamide, Paclitaxel, and Cisplatin (ITP) Chemotherapy (AG-ITP) in Patients With Metastatic or Locally Advanced Transitional Cell Carcinoma of the Urothelium
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic or Locally Advanced Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-095; CDR0000065841 (Registry Identifier: PDQ (Physician Data Query)); NCI-G97-1339
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter
Keywords: stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Filgrastim; Cisplatin; Doxorubicin; Gemcitabine; Ifosfamide; Paclitaxel

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: gemcitabine hydrochloride
Drug: ifosfamide
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy in treating patients with metastatic or locally advanced bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of doxorubicin, gemcitabine, and filgrastim (G-CSF) followed by ifosfamide, paclitaxel, cisplatin, and G-CSF in patients with metastatic or locally advanced transitional cell carcinoma of the urothelium.
* Determine the efficacy of this regimen in this patient population.

OUTLINE: This is a dose-escalation study of gemcitabine.

Patients receive doxorubicin IV over 30 minutes and gemcitabine IV on day 1 and filgrastim (G-CSF) subcutaneously (SC) on days 3-11. Treatment repeats every 2 weeks for 5 courses.

After completion of the fifth course, patients receive paclitaxel IV over 3 hours and cisplatin IV over 1 hour on day 1, ifosfamide IV over 1 hour on days 1-3, and G-CSF SC daily on days 6-17. Treatment repeats every 3-4 weeks for 4 courses.

Cohorts of 3-6 patients receive escalating doses of gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 3 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at the MTD.

PROJECTED ACCRUAL: A maximum of 20 patients will be accrued for phase I and a maximum of 10 patients will be accrued for phase II within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma of the urothelium
* Measurable disease, defined as unresectable or metastatic urothelial tract tumors OR
* Evaluable disease, defined as T3b or T4a bladder tumors

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count greater than 1,500/mm^3
* Platelet count greater than 150,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times normal
* SGOT less than 2 times normal

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* No serious cardiac arrhythmias, including first, second, or third degree heart block
* LVEF at least 50%

Other:

* No uncontrolled infection
* No other active malignancy except curatively treated nonmelanomatous skin cancer or carcinoma in situ of the cervix
* Fertile patients must use effective barrier contraception before, during, and for 6 months after study and are encouraged to continue for 2 years or longer after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1997-09; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean F. Bajorin, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Milowsky MI, Nanus DM, Maluf FC, Mironov S, Shi W, Iasonos A, Riches J, Regazzi A, Bajorin DF. Final results of sequential doxorubicin plus gemcitabine and ifosfamide, paclitaxel, and cisplatin chemotherapy in patients with metastatic or locally advanced transitional cell carcinoma of the urothelium. J Clin Oncol. 2009 Sep 1;27(25):4062-7. doi: 10.1200/JCO.2008.21.2241. Epub 2009 Jul 27. PMID 19636012